CLINICAL TRIAL: NCT00551031
Title: Immunogenicity and Safety of Two Dosages of the Split, Inactivated, Trivalent Influenza Vaccine Administered by Intradermal Route in the Elderly Compared With Standard Fluzone® in Adults and Elderly Subjects.
Brief Title: Study of Inactivated, Split-Virion Influenza Vaccine and Standard Fluzone® Vaccine in Adult and Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FID29
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Results first posted 2011-11-24 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Influenza; Myxovirus Infection
Keywords: Influenza; Orthomyxoviruses; Myxovirus Infection; Inactivated Split-virion influenza vaccine; Elderly
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Influenza Virus Vaccine Formulation 1 (Experimental): Influenza Virus Vaccine Formulation 1
  Interventions: Biological: Split, Inactivated, Trivalent Influenza Vaccine (Intradermal Formulation 1)
- Influenza Virus Vaccine Formulation 2 (Experimental): Influenza Virus Vaccine Formulation 2
  Interventions: Biological: Split, Inactivated, Trivalent Influenza Vaccine (Intradermal Formulation 2)
- Fluzone® Elderly Group (Active Comparator)
  Interventions: Biological: Split, Inactivated, Trivalent Influenza Vaccine (Standard dose)
- Fluzone® High-dose Group (Active Comparator): Participants enrolled at age ≥ 65 years
  Interventions: Biological: Split, Inactivated, Trivalent Influenza Vaccine (High-dose)
- Fluzone® Adults Group (Active Comparator): Participants enrolled at age 18-49 years.
  Interventions: Biological: Split, Inactivated, Trivalent Influenza Vaccine (Standard dose)

INTERVENTIONS:
Biological: Split, Inactivated, Trivalent Influenza Vaccine (Intradermal Formulation 1) — 0.1 mL, Intradermal (ID)
  Arms: Influenza Virus Vaccine Formulation 1
Biological: Split, Inactivated, Trivalent Influenza Vaccine (Intradermal Formulation 2) — 0.1 mL, Intradermal (ID)
  Arms: Influenza Virus Vaccine Formulation 2
Biological: Split, Inactivated, Trivalent Influenza Vaccine (Standard dose) — 0.5 mL, Intramuscular (IM)
  Other Names: Fluzone®
  Arms: Fluzone® Elderly Group
Biological: Split, Inactivated, Trivalent Influenza Vaccine (High-dose) — 0.5 mL, Intramuscular (IM)
  Other Names: Fluzone® High-dose
  Arms: Fluzone® High-dose Group
Biological: Split, Inactivated, Trivalent Influenza Vaccine (Standard dose) — 0.5 mL, Intramuscular (IM)
  Other Names: Fluzone®
  Arms: Fluzone® Adults Group

SUMMARY:
The present formulations are being developed for further study in the elderly population in order to generate additional supporting data.

Primary Objective:

To demonstrate non-inferiority of post-vaccination immunogenicity of subjects who received either 1 of the 2 investigational formulations of a trivalent inactivated vaccine (TIV) compared to that of the standard Fluzone® in elderly subjects.

Secondary Objectives:

Immunogenicity To describe the immunogenicity in subjects receiving investigational Fluzone and standard Fluzone®.

Safety:

To evaluate and describe the safety profile of investigational Fluzone in terms of solicited- and unsolicited adverse events and serious adverse events post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years or aged 18 to 49 years on the day of vaccination.
* Informed consent form signed.
* Medically stable (Subjects may have underlying illnesses such as hypertension, diabetes, ischemic heart disease or hypothyroidism, as long as their symptoms/signs are controlled. If they are on medication for a condition, the medication dose must have been stable for at least 3 weeks preceding vaccination.
* Able to attend all scheduled visits and to comply with all trial procedures.
* For a woman of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to vaccination, until at least 4 weeks after vaccination

Exclusion Criteria:

* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the standard-dose Fluzone® vaccine or to a vaccine containing any of the same substances.
* Known or suspected congenital or acquired immunodeficiency, hepatitis B (HBsAg) or hepatitis C infection or seropositivity immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* For a woman of child-bearing potential, known pregnancy or positive urine pregnancy test.
* Breast feeding woman.
* Neoplastic disease or any hematologic malignancy, (except localized skin or prostate cancer that is stable at the time of vaccination in the absence of therapy, as well as subjects who have a history of neoplastic disease and who have been disease free for ≥ 5 years).
* Current use of alcohol or recreational drugs that in the opinion of the Investigator may interfere with the subject's ability to comply with trial procedures.
* Receipt of blood or blood-derived products in the past 3 months that might interfere with the assessment of immune response.
* Vaccination against influenza in the past 6 months.
* Any vaccination in the 4 weeks preceding the trial vaccination.
* Planned receipt of any other vaccine in the four weeks following the trial vaccination.
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding trial vaccination.
* Planned participation in another clinical trial during the present trial period.

Note: Concomitant participation in an observational trial (not involving drugs, vaccines, or medical devices) is acceptable.

* Known thrombocytopenia or bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular vaccination.
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the investigator
* Personal or family history of Guillain-Barré Syndrome.
* Known current human immunodeficiency virus (HIV), hepatitis B (HBsAg) or hepatitis C infection or seropositivity.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* An acute febrile illness [oral temperature ≥ 99.5°F (≥ 37.5°C)] within 24 hours prior to vaccination. If this exists, vaccination will be deferred until the participant becomes afebrile.
* Signs and symptoms of an acute infectious respiratory illness. If this exists, vaccination will be deferred until the symptoms resolve.
* The use of an antibiotics therapy within 72 hours preceding the trial vaccination. If this exists, vaccination will be deferred until at least 72 hours after the last antibiotics therapy.
* Receipt of any allergy shots in the 7-day period prior to enrollment (vaccination), or scheduled to receive any allergy shots in the 7-day period after enrollment (vaccination). Subjects should be enrolled in the trial only if their allergy shots are given on a stable schedule outside the 7-day periods pre- and post-vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2098 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (29):
- United States (29):
  - Alabaster, Alabama
  - Mobile, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Fountain Valley, California
  - San Diego, California
  - Stanford, Connecticut
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Wichita, Kansas
  - Kansas City, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Allentown, Pennsylvania
  - Bensalem, Pennsylvania
  - Warwick, Rhode Island
  - Goose Creek, South Carolina
  - Fort Worth, Texas
  - Galveston, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Marshfield, Wisconsin

REFERENCES:
- [Derived] Tsang P, Gorse GJ, Strout CB, Sperling M, Greenberg DP, Ozol-Godfrey A, DiazGranados C, Landolfi V. Immunogenicity and safety of Fluzone((R)) intradermal and high-dose influenza vaccines in older adults >/=65 years of age: a randomized, controlled, phase II trial. Vaccine. 2014 May 1;32(21):2507-17. doi: 10.1016/j.vaccine.2013.09.074. Epub 2013 Oct 11. PMID 24120672
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 24 October to 31 October 2007 in 31 medical centers in the US.
Pre-assignment Details: A total of 2095 of the 2098 enrolled participants who met the inclusion and exclusion criteria were vaccinated.
Groups:
- Influenza Virus Vaccine Formulation 1: Participants aged 65 years or older who received 1 dose of Fluzone 15 µg intradermally (ID) using the Becton Dickenson Micro Injection System
- Influenza Virus Vaccine Formulation 2: Participants aged 65 years or older who received 1 dose of Fluzone 21 µg intradermally (ID) using the Becton Dickenson Micro Injection System
- Fluzone® Elderly Group: Participants aged 65 years or older who received 1 dose of Fluzone 15 µg intramuscularly (IM)
- Fluzone® High Dose Group: Participants aged 65 years or older who received 1 dose of Fluzone 60 µg intramuscularly (IM)
- Fluzone® Adults Group: Participants aged 18 to 49 years who received 1 dose of Fluzone 15 µg intramuscularly (IM)
Period: Overall Study
Arm/Group | Influenza Virus Vaccine Formulation 1 | Influenza Virus Vaccine Formulation 2 | Fluzone® Elderly Group | Fluzone® High Dose Group | Fluzone® Adults Group
Started | 637 | 636 | 319 | 320 | 186
Completed | 635 | 625 | 317 | 317 | 185
Not Completed | 2 | 11 | 2 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 1 | 2 | 0
Not completed — Serious Adverse Event | 0 | 2 | 1 | 0 | 0
Not completed — Did not receive vaccine | 1 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Virus Vaccine Formulation 1 | Influenza Virus Vaccine Formulation 2 | Fluzone® Elderly Group | Fluzone® High Dose Group | Fluzone® Adults Group | Total
Number analyzed (Participants) | 635 | 635 | 319 | 320 | 186 | 2095
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 186 | 186
  >=65 years | 635 | 635 | 319 | 320 | 0 | 1909
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.1 (6.03) | 72.9 (5.86) | 73.4 (5.91) | 73.0 (6.00) | 32.2 (8.49) | 64.8 (6.458)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 363 | 347 | 176 | 183 | 121 | 1190
  Male | 272 | 288 | 143 | 137 | 65 | 905
Region of Enrollment [Number; unit: Participants]
  United States | 635 | 635 | 319 | 320 | 186 | 2095

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) Before and After Vaccination With Fluzone Intradermal or Fluzone High Dose or Fluzone Intramuscular Vaccine.
Description: Serum antibody titers for the Influenza vaccine serogroups A/H1N1, A/H3N2, and B were assessed by hemagglutinin inhibition (HAI) assay.
Time Frame: Day 0 and Day 28 post vaccination
Population: Serum antibody titers GMTs were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influenza Virus Vaccine Formulation 1 | Influenza Virus Vaccine Formulation 2 | Fluzone® Elderly Group | Fluzone® High Dose Group | Fluzone® Adults Group
Number analyzed (Participants) | 607 | 608 | 304 | 309 | 179
Titers
  A/H1N1 Pre Dose (N=604, 607, 304, 309, 179) | 18.3 [16.9 to 19.8] | 18.6 [17.1 to 20.2] | 17.8 [15.7 to 20.0] | 17.3 [15.3 to 19.5] | 41.4 [32.6 to 52.7]
  A/H1N1 Post Dose (N=605, 607, 304, 309, 179) | 165.4 [149.2 to 183.4] | 174.1 [157.5 to 192.4] | 107.6 [93.2 to 124.3] | 236.1 [207.3 to 268.9] | 345.8 [294.1 to 406.6]
  A/H3N2 Pre Dose (N=606, 608, 304, 309, 179) | 103.8 [93.1 to 115.9] | 104.7 [93.9 to 116.7] | 95.1 [82.1 to 110.3] | 99.3 [84.6 to 116.7] | 73.0 [58.7 to 90.8]
  A/H3N2 Post Dose (N=605, 608, 304, 309, 179) | 348.3 [320.2 to 378.9] | 378.4 [346.9 to 412.7] | 276.9 [245.8 to 311.8] | 508.0 [452.6 to 570.1] | 398.3 [343.4 to 461.9]
  B Pre Dose (N=607, 608, 304, 309, 179) | 24.7 [22.9 to 26.6] | 25.1 [23.3 to 27.1] | 24.7 [22.2 to 27.4] | 24.1 [21.7 to 26.8] | 15.5 [13.4 to 17.9]
  B Post Dose (N=607, 608, 304, 309, 179) | 45.3 [42.3 to 48.4] | 47.5 [44.3 to 50.9] | 43.4 [39.2 to 48.0] | 59.9 [54.5 to 65.9] | 71.2 [61.7 to 82.3]

2. Primary Outcome: Percentage of Participants Who Achieved Seroconversion Post-Vaccination With Fluzone Intradermal or Fluzone High Dose or Fluzone Intramuscular Vaccine
Description: Seroconversion defined as either a pre-vaccination hemagglutination inhibition (HAI) titer < 1:10 and a post vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and a minimum four fold increase at one month post-vaccination.
Time Frame: Day 28 post-vaccination
Population: Serum antibody titers were assessed in the per protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Influenza Virus Vaccine Formulation 1 | Influenza Virus Vaccine Formulation 2 | Fluzone® Elderly Group | Fluzone® High Dose Group | Fluzone® Adults Group
Number analyzed (Participants) | 607 | 608 | 304 | 309 | 179
Percentage of Participants
  A/H1N1 (N=604, 607, 304, 309, 179) | 73 | 74 | 61 [0 to 0] | 82 | 62
  A/H3N2 (N=605, 608, 304, 309, 179) | 42 | 42 | 37 [0 to 0] | 56 | 52
  B (N=607, 608, 304, 309, 179) | 15 | 15 | 9 [0 to 0] | 26 | 44

3. Primary Outcome: Percentage of Participants Who Achieved Seroprotection Before and Post-vaccination With Fluzone Intradermal or Fluzone High Dose or Fluzone Intramuscular Vaccine.
Description: Seroprotection was defined as a Hemagglutination inhibition (HAI) titer ≥ 1:40
Time Frame: Day 0 and Day 28 post-vaccination
Population: Serum antibody titers were assessed in the per protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Influenza Virus Vaccine Formulation 1 | Influenza Virus Vaccine Formulation 2 | Fluzone® Elderly Group | Fluzone® High Dose Group | Fluzone® Adults Group
Number analyzed (Participants) | 607 | 608 | 304 | 309 | 179
Percentage of Participants
  A/H1N1 Pre Dose (N=604, 607, 304, 309, 179) | 27 | 25 | 25 | 23 | 49
  A/H1N1 Post Dose (N=605, 607, 304, 309, 179) | 88 | 90 | 79 | 94 | 97
  A/H3N2 Pre Dose (N=606, 608, 304, 309, 179) | 78 | 79 | 80 | 78 | 72
  A/H3N2 Post Dose (N=605, 608, 304, 309, 179) | 98 | 98 | 97 | 99 | 99
  B Pre Dose (N=607, 608, 304, 309, 179) | 38 | 37 | 39 | 37 | 25
  B Post Dose (N=607, 608, 304, 309, 179) | 65 | 67 | 62 | 77 | 79

4. Secondary Outcome: Number of Participants Reporting Solicited Injection Site or Systemic Reactions Post-vaccination With Either Fluzone Intradermal or Fluzone High Dose or Fluzone Intramuscular Vaccine.
Description: Solicited injection site reactions: Pain, Pruritus, Erythema, Swelling, Induration, and Ecchymosis.
  Solicited systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Chills
Time Frame: Days 0 through 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated subjects with available reaction data, intent to treat population.
Measure: Number; unit: Participants
Arm/Group | Influenza Virus Vaccine Formulation 1 | Influenza Virus Vaccine Formulation 2 | Fluzone® Elderly Group | Fluzone® High Dose Group | Fluzone® Adults Group
Number analyzed (Participants) | 635 | 635 | 319 | 320 | 186
Participants
  Any Injection Site Pain | 174 | 187 | 57 | 117 | 106
  Grade 3 Pain (Prevents daily activities) | 0 | 0 | 0 | 0 | 0
  Any Injection Site Pruritus | 204 | 214 | 27 | 17 | 24
  Grade 3 Pruritus (Prevents daily activities) | 2 | 3 | 0 | 0 | 0
  Any Injection Site Erythema | 426 | 434 | 48 | 55 | 29
  Grade 3 Erythema (≥ 5 cm) | 109 | 108 | 5 | 12 | 5
  Any Injection Site Swelling | 286 | 286 | 23 [0 to 0] | 45 | 14
  Grade 3 Swelling (≥ 5 cm) | 50 | 49 | 6 | 16 | 1
  Any Injection Site Induration | 310 | 311 | 33 | 45 | 20
  Grade 3 Induration (≥ 5 cm) | 41 | 43 | 5 | 12 | 4
  Any Injection Site Ecchymosis | 38 | 41 | 19 | 17 | 14
  Grade 3 Ecchymosis (≥ 5 cm) | 5 | 9 | 2 | 2 | 2
  Any Fever | 14 | 18 | 5 | 17 | 10
  Grade 3 Fever (> 102.2 ºF) | 0 | 0 | 0 | 0 | 1
  Any Headache | 103 | 89 | 41 | 59 | 61
  Grade 3 Headache (Prevents daily activities) | 2 | 6 | 1 | 2 | 2
  Any Malaise | 76 | 98 | 42 | 50 | 45
  Grade 3 Malaise (Prevents daily activities) | 5 | 3 | 0 [0 to 0] | 3 | 6
  Any Myalgia | 86 | 106 | 46 | 79 | 68
  Grade 3 Myalgia (Prevents daily activities) | 2 | 2 | 1 | 3 | 1
  Any Chills | 21 | 32 | 9 | 28 | 17
  Grade 3 Chills (Prevents daily activities) | 0 | 3 | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination up to 6 months post-vaccination.
Arm/Group | Influenza Virus Vaccine Formulation 1 | Influenza Virus Vaccine Formulation 2 | Fluzone® Elderly Group | Fluzone® High Dose Group | Fluzone® Adults Group
Serious Adverse Events (participants affected / at risk) | 34/635 | 38/635 | 21/319 | 16/320 | 7/186
Other Adverse Events (participants affected / at risk) | 426/635 | 434/635 | 57/319 | 117/320 | 106/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Influenza Virus Vaccine Formulation 1 (N=635) | Influenza Virus Vaccine Formulation 2 (N=635) | Fluzone® Elderly Group (N=319) | Fluzone® High Dose Group (N=320) | Fluzone® Adults Group (N=186)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1/319 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gasgtrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2/319 (2) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stent graft material failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Influenza Virus Vaccine Formulation 1 (N=635) | Influenza Virus Vaccine Formulation 2 (N=635) | Fluzone® Elderly Group (N=319) | Fluzone® High Dose Group (N=320) | Fluzone® Adults Group (N=186)
Injection site pain (General disorders) | 174 (174) | 187/632 (187) | 57 (57) | 117/318 (117) | 106/185 (106)
Injection site pruritus (General disorders) | 204 (204) | 214/632 (214) | 27 (27) | 17/318 (17) | 24/185 (24)
Injection site erythema (General disorders) | 426 (426) | 434/632 (434) | 48 (48) | 55/319 (55) | 29/185 (29)
Injection site swelling (General disorders) | 286 (286) | 286/631 (286) | 23 (23) | 45/319 (45) | 14/185 (14)
Injection site induration (General disorders) | 310 (310) | 311/631 (311) | 33 (33) | 45/319 (45) | 20/185 (20)
Injection site ecchymosis (General disorders) | 38/634 (38) | 41/631 (41) | 19 (19) | 17/319 (17) | 14/185 (14)
Fever (General disorders) | 14/630 (14) | 18/630 (18) | 5 (5) | 17/318 (17) | 10/182 (10)
Malaise (General disorders) | 76/634 (76) | 98/631 (98) | 42 (42) | 50/319 (50) | 45/185 (45)
Chills (General disorders) | 21/634 (21) | 32/632 (32) | 9 (9) | 28/319 (28) | 17/185 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 86/634 (86) | 106/632 (106) | 46 (46) | 79/319 (79) | 68/185 (68)
Headache (Nervous system disorders) | 103/634 (103) | 89/632 (89) | 41 (41) | 59/319 (59) | 61/185 (61)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.